CLINICAL TRIAL: NCT00092235
Title: Natural History Study of Clinical and Biological Factors Determining Outcomes in Chronic Graft-Versus-Host Disease
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Emory University, Department of Pediatrics (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040281; 04-C-0281; NCT00331968 (obsolete NCT alias)
Record Dates: First submitted 2004-09-21; First posted 2004-09-22 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12-11

CONDITIONS: Chronic Graft vs. Host Disease
Keywords: cGVHD-associated graft-versus-tumor effects (GVT); Allo-HSCT controls; Leukapheresis; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Patients who have undergone an allogeneic stem cell transplant and are diagnosed with cGVHD
- Cohort 2: Pediatric patients who have undergone an allogeneic stem cell transplant and are diagnosed with cGVHD
- Cohort 3: Patients who have undergone an allogeneic stem cell transplant and choose to submit biopsy, blood and urine samples only
- Cohort 4: Patients who have undergone an allogeneic stem cell transplant and are not diagnosed with cGVHD

SUMMARY:
Background:

* Chronic graft-versus-host disease (cGVHD) is a multi-organ alloimmune and autoimmune disorder that occurs following allogeneic hematopoietic stem cell transplantation (alloHSCT). It is characterized by immune dysregulation, immunodeficiency, impaired organ function, and decreased survival.
* Each year about 8000 patients receive allogeneic hematopoietic stem cell transplant (alloHSCT) in North America and about 50% of patients who are transplanted develop cGVHD.
* Chronic GVHD is also a disorder that simultaneously affects many organ systems in highly variable fashion and requires complex and coordinated medical management by multiple medical specialties. There is an urgent need for progress in understanding and effective treatments for cGVHD as it is one of the most serious complications of cancer therapy and hematopoietic stem cell transplantation.

Objectives:

* To establish a multidisciplinary clinic infrastructure for study of the pathogenesis and natural history of cGVHD.
* To prospectively identify clinical and biological prognostic markers in patients with cGVHD
* To develop clinically relevant cGVHD grading scales
* To identify novel biological characteristics of cGVHD and to describe them in the context of clinical history and presentation
* To identify potential clinical and biological markers of cGVHD activity
* To improve understanding of the biology of cGVHD-associated graft-versus-tumor effects
* To identify potential patients for cGVHD treatment protocols at the NCI and NIH

Eligibility:

-Patients age 1 and older referred by the primary transplant physician for the evaluation of chronic graft-versus-host disease independent of underlying diagnosis.

Design:

* Patient undergoes initial clinical and laboratory multispecialty work-up at the NCI cGVHD clinic.
* Minimally invasive biopsies and rarely, deep tissue biopsy may be obtained to confirm the diagnosis and/or rule-out other pathologic process (in adults only).
* Long tem data collection for evaluation of long-term outcomes will be conducted anually as feasible

DETAILED DESCRIPTION:
Background:

* Chronic graft-versus-host disease (cGVHD) is a multi-organ alloimmune and autoimmune disorder that occurs following allogeneic hematopoietic stem cell transplantation (alloHSCT). It is characterized by immune dysregulation, immunodeficiency, impaired organ function, and decreased survival.
* Each year about 8000 patients receive allogeneic hematopoietic stem cell transplant (alloHSCT) in North America and about 50% of patients who are transplanted develop cGVHD.
* Chronic GVHD is also a disorder that simultaneously affects many organ systems in highly variable fashion and requires complex and coordinated medical management by multiple medical specialties. There is an urgent need for progress in understanding and effective treatments for cGVHD as it is one of most serious complications of cancer therapy and hematopoietic stem cell transplantation.

Objectives:

* To establish a multidisciplinary clinic infrastructure for study of the pathogenesis and natural history of cGVHD
* To prospectively identify clinical and biological prognostic markers in patients with cGVHD
* To develop clinically relevant cGVHD grading scales
* To identify novel biological characteristics of cGVHD and to describe them in the context of clinical history and presentation
* To identify potential clinical and biological markers of cGVHD activity
* To improve understanding of the biology of cGVHD-associated graft-versus-tumor effects
* To identify potential patients for cGVHD treatment protocols at the NCI and NIH

Eligibility:

-Patients age 1 and older referred by the primary transplant physician for the evaluation of chronic graft-versus-host disease independent of underlying diagnosis.

Design:

* Patient undergoes initial clinical and laboratory multi-specialty work-up at the NCI cGVHD clinic
* Minimally invasive biopsies and rarely, deep tissue biopsy may be obtained to confirm the diagnosis and/or rule-out other pathologic process (in adults only)
* Long term data collection for evaluation of long-term outcomes will be conducted annually as feasible.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Any patient age 1 and older referred by the primary transplant physician for the evaluation of chronic graft-versus-host disease independently of age or underlying diagnosis
  2. Patient or the patient's legal representative is able and willing to provide consent.

EXCLUSION CRITERIA:

1. Significant medical condition or any other significant circumstance that could in the PIs assessment affect the patient's ability to tolerate, comply, or complete the study
2. Patients who in the PIs assessment have a life expectancy <3 months.

   Note: Because it is not always possible to make a clear clinical distinction between acute and chronic GVHD, patients with acute GVHD are not a-priori excluded until the possibility of chronic GVHD is reliably excluded on the basis of the clinical assessments in the cGVHD clinic.
3. Pregnant women are excluded from this study because multiple tests would need to be excluded for safety of the patient and the fetus.

Inclusion Criteria for control subjects without cGVHD:

* Age 1 and older
* Patient has undergone Allo-HSCT
* Patient or the patient's parent/guardian is able and willing to provide consent

Exclusion Criteria for control subjects without cGVHD:

* Active GVHD
* In the previous three months have received systemic immunosuppressant therapy for the treatment of GVHD
* In the previous three months have received therapy for malignancy

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected via referrals or from patients who were on companion clinical protocols at the NIH.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2004-10-26 (Actual)

PRIMARY OUTCOMES:
To prospectively identify candidate markers for clinical and biological prognostic factors in patients with cGVHD and develop a prognostic model | 2 years + 3 months after protocol entry
  Patient evaluations resulting in collection of data via several medical specialties; data will be examined individually and against clinical outcomes.
To improve our current understanding of the biology of cGVHD-associated graft-versus-tumor effects (GVT). | ongoing
  Studying mechanisms of how cGVHD exerts its anti-cancer effects via laboratory analysis.
To identify potential clinical and biological markers of cGVHD activity | ongoing
  Assessment of risk and outcome as related to molecular markers of pathogenesis and/or stage of disease.
To identify novel biological characteristics of cGVHD and to describe them in the context of clinical history and presentation | ongoing
  Through collection of data via several medical specialties, assess the weight of specific clinical and biological characteristics and disease severity scales for predicting major clinical outcomes.
To establish a multidisciplinary clinic infrastructure for study of pathogenesis and natural history of cGVHD | ongoing
  Assessment of clinical and biological characteristics of cGVHD.
To develop clinically relevant cGVHD grading scales | ongoing
  Develop appropriate staging as a tool for measuring responses or outcomes in clinical studies through prospective collection and analysis of data.

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Jurdi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the PI.@@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Zhao AT, Pirsl F, Steinberg SM, Holtzman NG, Schulz E, Mina A, Mays JW, Cowen EW, Comis LE, Joe GO, Yanovski JA, Pavletic SZ. Metabolic syndrome prevalence and impact on outcomes in patients with chronic graft-versus-host disease. Bone Marrow Transplant. 2023 Dec;58(12):1377-1383. doi: 10.1038/s41409-023-02097-y. Epub 2023 Sep 8. PMID 37684526
- [Derived] Schulz E, Pirsl F, Holtzman NG, Beshensky D, Cowen EW, Mitchell SA, Steinberg SM, Pavletic SZ. Red cell distribution width as a new prognostic biomarker in refractory chronic graft-versus-host disease. Haematologica. 2024 Jan 1;109(1):298-302. doi: 10.3324/haematol.2023.283646. No abstract available. PMID 37584292
- [Derived] Beshensky D, Pirsl F, Holtzman NG, Steinberg SM, Mays JW, Cowen EW, Comis LE, Joe GO, Magone MT, Schulz E, Waldman MA, Pavletic SZ. Predictors and significance of kidney dysfunction in patients with chronic graft-versus-host disease. Bone Marrow Transplant. 2023 Oct;58(10):1112-1120. doi: 10.1038/s41409-023-02032-1. Epub 2023 Jul 20. PMID 37474729
- [Derived] Yang AH, Han MAT, Samala N, Rizvi BS, Marchalik R, Etzion O, Wright EC, Cao L, Hakim FT, Jones E, Kapuria D, Hickstein DD, Fowler D, Kanakry JA, Kanakry CG, Kleiner DE, Koh C, Pavletic SZ, Heller T. Characterization of Hepatic Dysfunction in Subjects Diagnosed With Chronic GVHD by NIH Consensus Criteria. Transplant Cell Ther. 2022 Nov;28(11):747.e1-747.e10. doi: 10.1016/j.jtct.2022.07.017. Epub 2022 Jul 22. PMID 35878742
- [Derived] Ruben CL, Pirsl F, Steinberg SM, Holtzman NG, Parsons-Wandell L, Baruffaldi J, Curtis LM, Mitchell SA, Kerep AZ, Cowen EW, Berger A, Joe GO, Datiles MB 3rd, Mays JW, Pavletic SZ. Predictors of hematologic malignancy relapse in patients with advanced chronic graft-versus-host disease. Bone Marrow Transplant. 2021 Jul;56(7):1584-1592. doi: 10.1038/s41409-021-01211-2. Epub 2021 Feb 1. PMID 33526918
- [Derived] Katic M, Pirsl F, Steinberg SM, Dobbin M, Curtis LM, Pulanic D, Desnica L, Titarenko I, Pavletic SZ. Vitamin D levels and their associations with survival and major disease outcomes in a large cohort of patients with chronic graft-vs-host disease. Croat Med J. 2016 Jun 30;57(3):276-86. doi: 10.3325/cmj.2016.57.276. PMID 27374829
- [Derived] Curtis LM, Datiles MB 3rd, Steinberg SM, Mitchell SA, Bishop RJ, Cowen EW, Mays J, McCarty JM, Kuzmina Z, Pirsl F, Fowler DH, Gress RE, Pavletic SZ. Predictive models for ocular chronic graft-versus-host disease diagnosis and disease activity in transplant clinical practice. Haematologica. 2015 Sep;100(9):1228-36. doi: 10.3324/haematol.2015.124131. Epub 2015 Jun 18. PMID 26088932
- [Derived] Bassim CW, Fassil H, Dobbin M, Steinberg SM, Baird K, Cole K, Joe G, Comis LE, Mitchell SA, Grkovic L, Edwards D, Mays JW, Cowen EW, Pulanic D, Williams KM, Gress RE, Pavletic SZ. Malnutrition in patients with chronic GVHD. Bone Marrow Transplant. 2014 Oct;49(10):1300-6. doi: 10.1038/bmt.2014.145. Epub 2014 Jul 14. PMID 25029231
- [Derived] Martires KJ, Baird K, Steinberg SM, Grkovic L, Joe GO, Williams KM, Mitchell SA, Datiles M, Hakim FT, Pavletic SZ, Cowen EW. Sclerotic-type chronic GVHD of the skin: clinical risk factors, laboratory markers, and burden of disease. Blood. 2011 Oct 13;118(15):4250-7. doi: 10.1182/blood-2011-04-350249. Epub 2011 Jul 26. PMID 21791415
- [Derived] Clark J, Yao L, Pavletic SZ, Krumlauf M, Mitchell S, Turner ML, Cowen EW. Magnetic resonance imaging in sclerotic-type chronic graft-vs-host disease. Arch Dermatol. 2009 Aug;145(8):918-22. doi: 10.1001/archdermatol.2009.78. PMID 19687424
- [Derived] Imanguli MM, Swaim WD, League SC, Gress RE, Pavletic SZ, Hakim FT. Increased T-bet+ cytotoxic effectors and type I interferon-mediated processes in chronic graft-versus-host disease of the oral mucosa. Blood. 2009 Apr 9;113(15):3620-30. doi: 10.1182/blood-2008-07-168351. Epub 2009 Jan 23. PMID 19168793
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-C-0281.html